CLINICAL TRIAL: NCT04502381
Title: A Randomized Controlled Trial of Combined Inhalational With Intravenous Amphotericin B in Comparison With Intravenous Amphotericin B Alone for Treatment of Pulmonary Mucormycosis
Brief Title: Combined Inhalational With Intravenous Amphotericin B Versus Intravenous Amphotericin B Alone for Pulmonary Mucormycosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK/6146/DM/452
Record Dates: First submitted 2020-08-01; First posted 2020-08-06 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Mucormycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The study participants in the intervention arm will receive nebulization with amphotericin B deoxycholate (10 mg twice a day every alternate day, as described below) along with intravenous liposomal amphotericin B (3 to 5 mg/kg body weight)
  Interventions: Drug: Inhaled amp B deoxycholate+intravenous liposomal amp B; Drug: Intravenous liposomal amphotericin B alone
- Conventional arm (Active Comparator): Participants will receive treatment with only intravenous liposomal amphotericin B (3 to 5 mg/kg body weight)
  Interventions: Drug: Intravenous liposomal amphotericin B alone

INTERVENTIONS:
Drug: Inhaled amp B deoxycholate+intravenous liposomal amp B — Intravenous liposomal amphotericin B (beginning with 3mg/kg) along with inhaled amphotericin as below: Amp-B deoxycholate 50 mg (Amphotret™ Bharat serums and vaccines limited), will be dissolved in 10 mL distilled water. 2 mL of the reconstituted amphotericin B solution will be transferred into the drug chamber of a breath actuated nebulizer (Lupineb Ultra kit breath actuated nebulize which contains aeroclipse XL Reusable Breath Actuated Nebulizer and DeVilbiss 3655 compressor). 3 mL of distilled water is added to 2 mL of the reconstituted amphotericin B. The nebulization is continued till the chamber is emptied of the drug or the patient does not tolerate the therapy.
  The first three doses of amphotericin B nebulization will be under the direct supervision of a physician. If tolerated, nebulization will be continued twice a day till tolerated or till response.The patient will complete a VAS score for cough after nebulization.
  Arms: Intervention arm
Drug: Intravenous liposomal amphotericin B alone — Intravenous liposomal amphotericin B (beginning with 3mg/kg, up to 5 mg/kg), with or without surgery or other antifungals as clinically indicated

SUMMARY:
To assess the safety and feasibility of combined inhalational and intravenous amphotericin B therapy for the treatment of pulmonary mucormycosis. And compare the efficacy of combined therapy with that of intravenous amphotericin B alone.

DETAILED DESCRIPTION:
Pulmonary mucormycosis is a relatively a rare disease with a high mortality. The angioinvasion associated with mucormycosis prevents efficient drug delivery at the diseased site. Inhaled amphotericin B achieves drug levels in lung tissue and has been shown to be useful in several diseases including chronic pulmonary and allergic bronchopulmonary aspergillosis. Further inhaled forms of amphotericin B are associated with less nephrotoxicity and other systemic adverse effects. The role of inhaled amphotericin B in pulmonary mucormycosis has been previously demonstrated in murine models and anecdotal reports. The study hypothesis is that combined therapy with inhalational and intravenous amphotericin B is likely to result in better outcomes as compared with intravenous amphotericin B alone for treatment of pulmonary mucormycosis

ELIGIBILITY:
Inclusion Criteria:

Subjects with a clinicoradiologic suspicion of pulmonary mucormycosis will be enrolled if the diagnosis of mucormycosis is pathologically or microbiologically (smear showing aseptate hyphae, culture or molecular evidence showing Mucorales) confirmed. Cases of disseminated mucormycosis will be included, only if the pulmonary infection is confirmed pathologically or microbiologically from respiratory secretions or biopsy samples

Exclusion Criteria:

* Lack of informed consent
* Hypersensitivity to amphotericin B or any component of the formulation
* Pregnancy
* High likelihood of death within 48 h of enrolment
* Suspected pulmonary mucormycosis without histological or microbiologic proof

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Overall response (clinical and radiological improvement) at the end of six weeks of start of therapy | 6 weeks after the start of therapy
  Complete response: Survival and resolution of all attributable symptoms and signs of disease plus Resolution of radiological lesion(s); persistence of only a scar or postoperative changes can be equated with complete radiological response Partial response: Survival and improvement of attributable symptoms and signs of disease plus At least 25% reduction in diameter of radiological lesion OR In cases of radiological stabilization (defined as 0%-25% reduction in the diameter), resolution of all attributable symptoms and signs of fungal disease can be equated with a partial response Stable response: Survival and minor or no improvement in attributable symptoms and signs; plus Radiological stabilization (defined as 0%-25% reduction in diameter) Progression: Worsening clinical symptoms or signs plus New sites of disease or radiological worsening Death Complete and partial response will be called "success"
Adverse events related to therapy | till 6 weeks from randomization (start of therapy)
  Adverse events related to therapy (especially, incidence of bronchospasm and acute kidney injury)

SECONDARY OUTCOMES:
In-hospital mortality | During hospital stay, approximately till 6 weeks from randomization (start of therapy)
  Death due to any cause in-hospital
90 day mortality | 90 days from the date of randomization
  Death due to any cause till 90 days of randomization
Proportion of subjects requiring discontinuation or modification of therapy due to adverse events | till 6 weeks from randomization (start of therapy)
  Number of participants withdrawing therapy in each arm, divided by the total number of patients in the same arm

CONTACTS AND LOCATIONS:
Overall Officials: Ratnakara Rao, MBBS, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post graduate Institute medical education and research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No